CLINICAL TRIAL: NCT06516146
Title: Impact 360 Study for Healthy Agers
Brief Title: Impact 360 for Healthy Agers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: The Jack and Darlene Poole Foundation (Unknown)
Responsible Party: Principal Investigator, Silke Cresswell, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H21-01750
Record Dates: First submitted 2024-05-03; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Healthy Aging
Keywords: Exercise; Mindfulness; Microbiome; Well-Being
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Meditation; Diet

STUDY DESIGN:
Intervention Model Description: Adults 50-75 years of age without a diagnosis of a neurodegenerative condition, will be recruited and screened for eligibility. Sixty participants will be randomly assigned to the waitlist group or the intervention group and will be striated into cohorts blocks. Each cohort block will start the intervention at the same time and will participate in the intervention together. This will allow for social interaction, engagement with their peers, and hopefully encouraging better adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise, Diet, Mindfulness (Experimental): The intervention group will start the intervention immediately following their baseline assessment. They will undergo another assessment after the 6 month intervention period.
  Interventions: Behavioral: Exercise; Behavioral: Meditation; Behavioral: Diet
- Waitlist Group (No Intervention): Participants randomized into the waitlist group will undergo a baseline assessment, and will then be encouraged to continue their daily activities as usual for 6 months. Physical activity and sleep will be monitored during this time using wearable devices. Links to questionnaires will be emailed monthly. After the 6-month waitlist period, participants will undergo a second assessment prior to starting the intervention. The multimodal intervention will be 6-months in length, using the same measures of adherence, and will be followed by a final assessment.

INTERVENTIONS:
Behavioral: Exercise — The intervention will involve online (via University of British Colombia (UBC) Zoom videoconferencing) 1-hour moderate to high intensity exercise classes 3 times a week for 6 months
  Arms: Exercise, Diet, Mindfulness
Behavioral: Meditation — The intervention will involve 15 minute guided mediation following exercise classes as well as mindfulness classes.
  Mindfulness classes will consist of 1.5 hour Mindfulness Based Stress Reduction (MBSR) classes for the first 2 months, followed by 1 month of 1 hour bi-weekly discussions and practice, then MBSR 2.0 for months 4 and 5, and 1 hour bi-weekly discussions and practice for the remaining month of the intervention.
  Arms: Exercise, Diet, Mindfulness
Behavioral: Diet — The intervention will involve biweekly 1-hour nutrition and cooking classes with a dietician.
  Arms: Exercise, Diet, Mindfulness

SUMMARY:
The Impact 360 study will evaluate the effects of a combined intervention of exercise, mindfulness, and nutrition on 8 key indicators of health and the mechanisms that drive these changes. 60 subjects aged 50 to 75 without a current diagnosis of a brain disorder will be recruited. This study will follow a partial crossover design. All participants will receive the intervention. Participants randomized into the intervention group after their baseline screening will receive the 6-month intervention. Those randomized into the waitlist group will complete another assessment at the end of the 6-month care as usual phase before receiving the intervention.

DETAILED DESCRIPTION:
Current research suggests that exercise, meditation, and nutrition have neuroprotective effects although there is still a lack of pharmacological therapies to prevent or slow down disease progression. The benefits of these individual interventions have been shown, but emerging evidence suggests that combined interventions are more powerful than isolated ones. The crucial next step is to study the impact of a multimodal program on brain health and to comprehensively examine underlying mechanisms.

The comprehensive assessment ("360 degree approach") will focus on 8 key areas of health: cognition, inflammation, microbiome diversity, sleep quality, neurological imaging markers, physical fitness, cardiovascular health, and social and mental well-being. This comprehensive assessment in this healthy aging cohort will serve two purposes: 1) Help us to understand the mechanisms behind the benefits of this multimodal intervention and how the interactive effects influence one's overall health and 2) to serve as a normative dataset for replication of this study in clinical populations (e.g. Parkinson's disease, Alzheimer's disease, stroke)

The objective of this study is to explore the effects of this combined intervention on overall health. The investigators aim to discover the mechanisms of action behind the benefits of this multimodal intervention. The investigators will assess the impact of the intervention on overall health using the following 8 key indicators of overall health: cognition, inflammation and biomarkers, gut microbiome diversity, sleep quality, Magnetic Resonance Imaging (MRI) neurological markers, cardiorespiratory fitness and physical health, cardiovascular disease risk factors, and emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are able to complete questionnaires and follow directions for interventions
* Have access to a smartphone that can support the Fitbit app

Exclusion Criteria:

* Any neurological disease/disorder diagnosis (Ex: Parkinson's Disease, Multiple Sclerosis, Traumatic Brain Injury, Brain lesion, Stroke, etc)
* Any chronic medical condition which would affect ability to participate in exercise
* Any contraindication for exercise based on the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) and medical clearance form
* Participants who were told by a medical doctor that they need to be medically supervised for exercise
* Montreal Cognitive Assessment (MoCA) scores <21/30
* Significant cognitive impairment, depression, or eating disorder
* Any contraindication to MRI scanning; such as implanted metal clips or wires (see list below)
* Participants currently doing 180 minutes or more of moderate-vigorous intensity exercise per week AND either of the following:
* Completion of an Mindfulness-Based Stress Reduction course OR; Score >8/15 in the Mediterranean-Dietary Approaches to Stop Hypertension (DASH) Intervention for Neurodegenerative Delay (MIND) Diet Questionnaire
* Significant or unstable cardiovascular or respiratory disease
* Severe/multiple head trauma(s)
* Subjects who are pregnant or breastfeeding
* Subjects with a history or major episodes of drug or alcohol abuse
* Chronic/acute bacterial/viral infection
* GI cancer
* Inflammatory bowel disease

Exclusion for MRI scanning:

* Individuals weighing > 400 lbs (limit of MRI machine)
* Artificial heart valve
* Brain aneurysm clip
* Electrical stimulator for nerves or bones
* Ear or eye implant
* Implanted drug infusion pump
* Coil, catheter, or filter in any blood vessel
* Orthopedic hardware (artificial joint, plate, screws)
* Other metallic prostheses
* Shrapnel, bullets, or other metal fragments
* Surgery or tattoos (including tattooed eyeliner) in the last six weeks
* Brain surgery
* Have a cardiac pacemaker, wires or defibrillator
* Have had an injury where a piece of metal lodged in the eye or orbit
* Have a ferromagnetic aneurysm clip

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-01-05 (Estimated); Study Completion 2025-01-05 (Estimated)

PRIMARY OUTCOMES:
Cognition - NIH Toolbox Cognitive Battery | 6 Months
  Cognition will be measured using the National Institutes of Health (NIH) Toolbox Cognitive battery (NIHTB-CB). Testing is done pre- and post-intervention to compare scores.
Cognition- Montreal Cognitive Assessment | 6 Months
  Cognition will be measured using the Montreal Cognitive Assessment (MoCA). Testing is done pre- and post-intervention to compare scores.
Cognition- Parkinson's Disease Cognitive Rating Scale | 6 Months
  Cognition will be measured using the Parkinson's Disease Cognitive Rating Scale (PD-CRS). Testing is done pre- and post-intervention to compare scores.
Inflammation and Biomarkers in Serum- High Sensitivity C-Reactive Protein | 6 Months
  Systemic inflammation will be assessed by measuring concentrations of high sensitivity C-reactive protein (hs-CRP). Samples will be taken pre- and post-intervention to assess changes.
Inflammation and Biomarkers in Serum - Interleukin-1β | 6 Months
  Systemic inflammation will be assessed by measuring concentrations of interleukin-1β (IL-1β). Samples will be taken pre- and post-intervention to assess changes.
Inflammation and Biomarkers in Serum - Interleukin-6 | 6 Months
  Systemic inflammation will be assessed by measuring concentrations of interleukin-6 (IL-6). Samples will be taken pre- and post-intervention to assess changes.
Inflammation and Biomarkers in Serum - Tumour Necrosis Factor Alpha | 6 Months
  Systemic inflammation will be assessed by measuring concentrations of Tumour Necrosis Factor Alpha (TNFa). Samples will be taken pre- and post-intervention to assess changes.
Inflammation and Biomarkers in Serum - Interleukin-8 | 6 Months
  Systemic inflammation will be assessed by measuring concentrations of interleukin-8 (IL-8). Samples will be taken pre- and post-intervention to assess changes.
Inflammation and Biomarkers in Serum - Interleukin-10 | 6 Months
  Systemic inflammation will be assessed by measuring concentrations of interleukin-10 (IL-10). Samples will be taken pre- and post-intervention to assess changes.
Inflammation and Biomarkers in Serum - Interleukin-18 | 6 Months
  Systemic inflammation will be assessed by measuring concentrations of interleukin-18 (IL-18). Samples will be taken pre- and post-intervention to assess changes.
Inflammation and Biomarkers in Serum - Calprotectin | 6 Months
  Systemic inflammation will be assessed by measuring concentrations of calprotectin. Samples will be taken pre- and post-intervention to assess changes.
Inflammation and Biomarkers in Serum - cortisol | 6 Months
  Systemic inflammation will be assessed by measuring concentrations of cortisol. Samples will be taken pre- and post-intervention to assess changes.
Microbiome Diversity | 6 Months
  Stool samples will be analyzed for gut microbiome composition by shallow shotgun metagenome sequencing. Samples will be taken pre- and post-intervention to assess changes.
Sleep Efficiency | 6 Months
  Sleep efficiency (total sleep time/time spent in bed) will be measured through a wearable device with an accelerometer. This device will also measure other components of sleep quality such as sleep onset latency, total sleep time and wake after sleep onset.
Pittsburgh Sleep Quality Index | 6 Months
  The Pittsburgh Sleep Quality Index will be used to collect subjective sleep quality data on a monthly basis.
Total Grey Matter Volume | 6 Months
  Total grey matter volume will be measured using an MRI. Testing is done pre- and post-intervention to compares scores.
Hippocampal Volume | 6 Months
  Hippocampal volume will be measured using an MRI. Testing is done pre- and post-intervention to compares scores.
White matter hyperintensities volume | 6 Months
  White matter hyperintensities volume will be measured using an MRI. Testing is done pre- and post-intervention to compares scores.
Myelin Water | 6 Months
  Myelin water imaging will be collected using resting state functional MRI. Testing is done pre- and post-intervention to compares scores.
Functional MRI | 6 Months
  A flanker task will be administered during the MRI to examine selective attention, inhibitory function, and executive control. Testing is done pre- and post-intervention to compares scores.
Maximal oxygen consumption (VO2 Max) | 6 Months
  Predicted maximal oxygen consumption will be measured using a six-minute walk test. Testing is done pre- and post-intervention to compares scores.
Heart Rate Recovery | 6 Months
  Heart rate recovery will be measured using a three-minute step test. Testing is done pre- and post-intervention to compares scores.
Berg Balance Assessment | 6 Months
  A Berg Balance Assessment will be used to measure participants balance. Testing is done pre- and post-intervention to compares scores.
Dynamic Gate Index | 6 Months
  The Dynamic Gait Index will be used to measure participants gait. Testing is done pre- and post-intervention to compares scores.
Timed Up and Go Test | 6 Months
  The Dynamic Gait Index will be used to measure participants gait. Testing is done pre- and post-intervention to compares scores.
30 Second Sit to Stand Test | 6 Months
  Functional lower extremity strength with be assessed using the 30 second sit to stand test. Testing is done pre- and post-intervention to compare scores.
Dual-Energy X-Ray Absorptiometry (DEXA) | 6-Months
  Body composition, such as body fat and muscle mass, will be measured using Dual-energy X-ray Absorptiometry. Testing is done pre- and post-intervention to compare scores.
Physical Activity Levels | 6 Months
  Physical activity levels will be measured through a wearable device to help ensure adherence and effectiveness of the exercise intervention. Data will be collected throughout the study.
Heart Rate | 6 Months
  Heart rate will be measured through a wearable device to help ensure adherence and effectiveness of the exercise intervention. Data will be collected throughout the study.
Fried Frailty Index | 6 Months
  Physical frailty will be assessed using the fried frailty index. Testing is done pre- and post-intervention to compares scores.
Blood Pressure | 6 Months
  Blood pressure will be measured pre- and post-intervention to compares scores.
Weight | 6 Months
  Weight will be measured pre- and post-intervention to compares scores.
Framingham Risk Score | 6 Months
  Cardiovascular health will be assessed using the Framingham Risk Score. This score includes measurements of age, total cholesterol, smoking status, HDL level, diabetes status, systolic blood pressure and treatment status. Testing is done pre- and post-intervention to compares scores.
NIH Toolbox- Emotional Battery | 6 Months
  Social, emotional, and mental well-being will be evaluated using the NIH Toolbox-Emotional Battery. Testing is done pre- and post-intervention to compares scores.
World Health Organization (WHO) Quality of Life Questionnaire | 6 Months
  Quality of life will be evaluated using the World Health Organization (WHO) Quality of Life Questionnaire. Testing is done pre- and post-intervention to compares scores.
Freiburg Mindfulness Inventory | 6 Months
  Questionnaires related to mindfulness will be administered throughout the study at monthly intervals.
Mindful Attention Awareness Scale | 6 Months
  Questionnaires related to mindfulness will be administered throughout the study at monthly intervals.
Multidimensional Assessment of Interoceptive Awareness | 6 Months
  Questionnaires related to mindfulness will be administered throughout the study at monthly intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Silke Appel-Cresswell, MD, FRCPC, Principal Investigator — University of British Colombia
Locations (1):
- University of British Colombia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No